CLINICAL TRIAL: NCT04118803
Title: Observational Study on Inappropriate Therapies After Replacement of ICDs
Brief Title: Observational Study on Inappropriate Therapies
Acronym: OSIRIS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Other Study IDs: RTSY04 - OSIRIS
Record Dates: First submitted 2019-10-05; First posted 2019-10-08 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Inappropriate Shocks From Implanted Defibrillator; ICD Replacement or Upgrade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ICD replacement or upgrade — Currently, it is common for patients to survive beyond their initial prophylactic ICD generator. It is unclear whether further benefit related to inappropriate shocks or ATP is derived from long-term device therapy, particularly if there has been a change in the patient's cardiovascular condition.

SUMMARY:
The purpose of the study is to assess the incidence of inappropriate shocks at 2 years, in a population of patients undergoing a generator replacement (VR/DR/CRT) or upgrade from a previously implanted ICD (VR/DR)

DETAILED DESCRIPTION:
All subjects will be included during an inclusion visit (within 7 days post generator replacement or upgrade), and followed up at a post replacement visit (1 - 6 months post replacement or upgrade), at 12, 18 and 24 months post replacement or upgrade. These follow-up visits will be performed in-clinic except for the 18 months post replacement or upgrade visit, which could be performed through device remote monitoring.

Additional follow-ups can be performed at physician's discretion. Data on reportable adverse events will be collected throughout the study. All study data will be collected using an EDC system.

All delivered anti-tachycardia therapies (shock or ATP) will be reviewed by an independent board of experts in order to evaluate appropriateness.

The programming of the device parameters is at physician's discretion (suggested settings is slow VT monitoring zone 150 - 185 bpm with 30 cycles persistence, VT zone 185 - 230 bpm with 16 cycles persistence, remote monitoring activated).

ELIGIBILITY:
Inclusion Criteria:

1. Any subject that had an ICD/CRT-D replacement/upgrade according to the latest relevant clinical guidelines with a MicroPort CRM ICD / CRT-D for less than 7 days
2. Signed and dated the informed consent form

Exclusion Criteria:

1. RV lead replacement
2. Previous ICD/CRT-D inactivated or already explanted
3. Active myocarditis
4. Primary prevention for Arrhythmogenic Ventricular Cardiomyopathy, Ion channelopathies, Hypertrophic Cardiomyopathy and Infiltrative or Inherited Cardiomyopathy.
5. Heart transplant (done or on waiting list) or implanted with a ventricular assist device (VAD)
6. Already included in an Interventional study that could confound the results of this study
7. Inability to understand the purpose of the study or to meet follow-up visits as defined in the investigational plan
8. Minor age (<18 years) or under guardianship or kept in detention
9. Ongoing drug or alcohol addiction or abuse which would interfere with the subject's ability to be compliant with the study.
10. Life expectancy less than 1 year
11. Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for an ICD or CRT-D implant according to the latest applicable guidelines and requiring a device replacement or system upgrade from a previous ICD (VR/DR/CRT-D).
Sampling Method: Probability Sample
Enrollment: 881 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of inappropriate shocks | 2 years after replacement or upgrade
  This endpoint will assess the incidence of inappropriate shocks, in a population of patients undergoing a generator replacement (VR/DR/CRT) or upgrade from a previously implanted ICD (VR/DR).

CONTACTS AND LOCATIONS:
Overall Officials: Christoff Kolb, Dr., Principal Investigator — Deutsches Herzzentrum, Lazarettstraße 36, 80636 Munich, Germany
Locations (58):
- United States (5):
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - The University of Chicago Medicine Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - St. Mary Medical Center, Langhorne, Pennsylvania
- Austria (3):
  - Universitätsklinik Innsbruck - Kardiologie und Angiologie, Innsbruck
  - Akademisches Krankenhaus Wien, Vienna
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Belgium (2):
  - UZ Brussel, Jette
  - UCL Mont-Godinne, Yvoir
- France (19):
  - CH du Pays d'Aix, Aix-en-Provence
  - CH Annecy Genevois, Annecy
  - Clinique Rhône Durance, Avignon
  - CHU Brest, Brest
  - Hôpital d'Instruction des Armées Percy, Clamart
  - CHU de Grenoble, Grenoble
  - CH de Libourne Robert Boulin, Libourne
  - CHU Dupuytren, Limoges
  - Hôpital Nord, Marseille
  - Hôpital Privé Clairval, Marseille
  - Clinique du Millénaire, Montpellier
  - CHU Nice, Nice
  - CHU Groupe HU Caremeau, Nîmes
  - CH de Perpignan CHG St Jean, Perpignan
  - CHU Poitiers, Poitiers
  - CHU - Hôpital Nord - Saint-Étienne, Saint-Etienne
  - CHI Toulon La Seyne Sur Mer, Toulon
  - Centre Hospitalier de Rangueil, Toulouse
  - Centre Hospitalier de Valence, Valence
- Germany (4):
  - UKSH Schleswig Holstein Campus Kiel, Kiel
  - Deutsches Herzzentrum München, Munich
  - Cardiologicum, Pirna
  - Katharinen Hospital Unna, Unna
- Italy (12):
  - Ospedale L. Bonomo, Andria
  - Azienda Ospedaliera G. Moscati, Avellino
  - Ospedale Clinicizzato SS. Annunziata, Chieti
  - Presidio Ospedaliero di Chioggia, Chioggia
  - Ospedale Santa Maria dei Battuti, Conegliano
  - Ospedale San Salvatore, L’Aquila
  - Grande Ospedale Metropolitano Niguarda Ca Granda, Milan
  - Ospedale S. Gerardo, Monza
  - Ospedale Policlinico Federico II, Napoli
  - Ospedale Giovanni Paolo II, Ragusa
  - Ospedale Giuseppe Mazzini, Teramo
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Di Trieste, Trieste
- Isala Klinieken, Zwolle, Netherlands
- Centro Hospitalar Lisboa Norte - Hospital de Santa Maria, Lisbon, Portugal
- Spain (6):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de La Ribera, Alzira
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario de Valencia, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - GZO Spital Wetzikon AG, Wetzikon
- United Kingdom (3):
  - Belfast Health & Social Care Trust, Belfast
  - Papworth Hospital NHS Foundation Trust, Cambridge
  - Northampton General Hospital NHS TRUST, Northampton

IPD SHARING:
Plan to Share IPD: No
A clinical study report will be completed at the end of the study and publication of study results may be performed